CLINICAL TRIAL: NCT02490384
Title: Randomized Control Trial Physical Exam Indicated Cerclage in Twin Gestations
Brief Title: Physical Exam Indicated Cerclage in Twin Gestations
Acronym: TWIN-PEIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to significant decrease of perinatal mortality in the cerclage group
Sponsor: Thomas Jefferson University (Other)
Collaborators: Columbia University (Other); Federico II University (Other); Albany Medical College (Other); University of Rochester (Other); George Washington University (Other); Wright State University (Other); Baystate Medical Center (Other); Università degli Studi di Brescia (Other); University of Bologna (Other); University Hospital, Geneva (Other); University of Warsaw (Other); Maternal Fetal Medicine Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ThomasJeffersonU
Record Dates: First submitted 2015-06-29; First posted 2015-07-03 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Twin Pregnancy, Antepartum Condition or Complication; Preterm Birth; Cervical Dilation Premature
Keywords: Cervical cerclage
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical exam indicated cerclage (Active Comparator): Cerclage
  Interventions: Procedure: Physical exam indicated cerclage
- Expectant management (No Intervention): No cerclage

INTERVENTIONS:
Procedure: Physical exam indicated cerclage — Cervical cerclage
  Arms: Physical exam indicated cerclage

SUMMARY:
This is a multicenter randomized study designed to determine if physical exam indicated cerclage reduces the incidence of spontaneous preterm birth <34 weeks in asymptomatic women with twin gestations and dilated cervix, diagnosed by pelvic exam between 16 to 23 6/7 weeks of gestation.

DETAILED DESCRIPTION:
Twin pregnancies have 58% incidence of preterm delivery (before 37 weeks of gestation), with increased perinatal mortality and neonatal morbidity. No therapy has proven effective in preventing preterm birth in twins. When cervical dilation is identified before 24 weeks in singleton pregnancies, the risk of preterm birth is 90%-100%; based on a small series of cases, approximately 50% of twin gestations with cervical dilation will be delivered prior to viability (24 weeks) and the risk of preterm birth prior to 34 and 37 weeks was 85% and 100%. Cervical dilation is the worst prognostic factor for preterm birth. There are a small number of case reports of cervical cerclage in twin pregnancies with a dilated cervix that suggest similar outcomes to those in singleton pregnancies. The investigators' objective is to determine if physical exam indicated cerclage reduces the incidence of spontaneous preterm birth <34 weeks and improve perinatal outcome in asymptomatic women with twin gestations and dilated cervix (1 to 5 cm) between 16 to 23 6/7 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women older than 18 years of age
2. Diamniotic twin pregnancy
3. Cervical dilation between 1 to 5 cm and/or visible membranes by pelvic exam or speculum exam between at 16-23 6/7 weeks gestation

Exclusion Criteria:

1. Singleton pregnancy or higher order than twins multiple gestation
2. Cervical dilation more than 5 cm
3. Amniotic membranes prolapsed beyond external os into the vagina, unable to visualize cervical tissue
4. More than 24 weeks of gestation
5. Multifetal reduction after 14 weeks
6. Monoamniotic twins
7. Twin-twin transfusion syndrome
8. Ruptured amniotic membranes at the time of diagnosis of dilated cervix
9. Major fetal structural anomaly
10. Fetal chromosomal abnormality
11. Cerclage already in place for other indications
12. Active vaginal bleeding
13. Suspicion of clinical or biochemical chorioamnionitis
14. Painful regular uterine contractions
15. Labor (progressing cervical dilation)
16. Placenta previa

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Preterm delivery less than 34 weeks | at delivery
  Incidence of preterm birth less than 34 weeks (any indication)

SECONDARY OUTCOMES:
Spontaneous preterm birth less than 34 | at delivery
  Incidence of spontaneous preterm birth less than 34 weeks
Preterm delivery less than <32 weeks, <28 weeks, or <24 weeks | at delivery
  Incidence of preterm birth less than <32 weeks, <28 weeks, or <24 weeks
Mean gestational age at delivery | at delivery
  Mean value of gestational age at delivery (weeks)
Birth weight at birth | at delivery
  Mean value (grams)
Gestational age at spontaneous rupture of membranes | at presentation of rupture membranes
  Mean value (weeks) through study completion

OTHER OUTCOMES:
Chorioamnionitis | Time of delivery
  Incidence
Composite adverse neonatal outcome | Incidence between birth and 28 days of age
  Includes necrotizing enterocolitis, intraventricular hemorrhage (grade 3 or higher), respiratory distress syndrome, bronchopulmonary dysplasia, retinopathy, blood-culture proven sepsis
Fetal demise | Incidence before delivery
  Incidence
Neonatal death | Incidence between birth and 28 days of age
  Incidence
Perinatal death | Incidence before and after birth ulntil 28 days of age
  Incidence
Maternal death | Between birth and 6 weeks postpartum
  Incidence
Interval between diagnosis and delivery | at delivery
  Mean value (days) through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Roman, MD, Principal Investigator — amanda.roman@jefferson.edu
Locations (11):
- United States (7):
  - George Washington University, Washington D.C., District of Columbia
  - Albany Medical Center, Albany, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wright State University, Dayton, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Austin Maternal Fetal Medicine St David's Health Care, Austin, Texas
- Italy (3):
  - Bologna University, Bologna
  - University of Brescia, Brescia
  - Università degli Studi di Napoli "Federico II", Naples
- University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
De identified data
Supporting Information: Study Protocol, SAP, CSR
Time Frame: June 2020 2 years
Access Criteria: x

REFERENCES:
- [Background] Hamilton BE, Hoyert DL, Martin JA, Strobino DM, Guyer B. Annual summary of vital statistics: 2010-2011. Pediatrics. 2013 Mar;131(3):548-58. doi: 10.1542/peds.2012-3769. Epub 2013 Feb 11. PMID 23400611
- [Background] Goldenberg RL, Iams JD, Miodovnik M, Van Dorsten JP, Thurnau G, Bottoms S, Mercer BM, Meis PJ, Moawad AH, Das A, Caritis SN, McNellis D. The preterm prediction study: risk factors in twin gestations. National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Am J Obstet Gynecol. 1996 Oct;175(4 Pt 1):1047-53. doi: 10.1016/s0002-9378(96)80051-2. PMID 8885774
- [Background] Conde-Agudelo A, Romero R, Hassan SS, Yeo L. Transvaginal sonographic cervical length for the prediction of spontaneous preterm birth in twin pregnancies: a systematic review and metaanalysis. Am J Obstet Gynecol. 2010 Aug;203(2):128.e1-12. doi: 10.1016/j.ajog.2010.02.064. Epub 2010 Jun 23. PMID 20576253
- [Background] Rouse DJ, Caritis SN, Peaceman AM, Sciscione A, Thom EA, Spong CY, Varner M, Malone F, Iams JD, Mercer BM, Thorp J, Sorokin Y, Carpenter M, Lo J, Ramin S, Harper M, Anderson G; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A trial of 17 alpha-hydroxyprogesterone caproate to prevent prematurity in twins. N Engl J Med. 2007 Aug 2;357(5):454-61. doi: 10.1056/NEJMoa070641. PMID 17671253
- [Background] Schuit E, Stock S, Groenwold RH, Maurel K, Combs CA, Garite T, Spong CY, Thom EA, Rouse DJ, Caritis SN, Saade GR, Zachary JM, Norman JE, Rode L, Klein K, Tabor A, Cetingoz E, Morrison JC, Magann EF, Briery CM, Serra V, Perales A, Meseguer J, Nassar AH, Lim AC, Moons KG, Kwee A, Mol BW. Progestogens to prevent preterm birth in twin pregnancies: an individual participant data meta-analysis of randomized trials. BMC Pregnancy Childbirth. 2012 Mar 15;12:13. doi: 10.1186/1471-2393-12-13. PMID 22420582
- [Background] Romero R, Nicolaides K, Conde-Agudelo A, Tabor A, O'Brien JM, Cetingoz E, Da Fonseca E, Creasy GW, Klein K, Rode L, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone in women with an asymptomatic sonographic short cervix in the midtrimester decreases preterm delivery and neonatal morbidity: a systematic review and metaanalysis of individual patient data. Am J Obstet Gynecol. 2012 Feb;206(2):124.e1-19. doi: 10.1016/j.ajog.2011.12.003. Epub 2011 Dec 11. PMID 22284156
- [Background] Saccone G, Rust O, Althuisius S, Roman A, Berghella V. Cerclage for short cervix in twin pregnancies: systematic review and meta-analysis of randomized trials using individual patient-level data. Acta Obstet Gynecol Scand. 2015 Apr;94(4):352-8. doi: 10.1111/aogs.12600. Epub 2015 Mar 1. PMID 25644964
- [Background] Roman A, Rochelson B, Fox NS, Hoffman M, Berghella V, Patel V, Calluzzo I, Saccone G, Fleischer A. Efficacy of ultrasound-indicated cerclage in twin pregnancies. Am J Obstet Gynecol. 2015 Jun;212(6):788.e1-6. doi: 10.1016/j.ajog.2015.01.031. Epub 2015 Jan 28. PMID 25637840
- [Background] Rebarber A, Bender S, Silverstein M, Saltzman DH, Klauser CK, Fox NS. Outcomes of emergency or physical examination-indicated cerclage in twin pregnancies compared to singleton pregnancies. Eur J Obstet Gynecol Reprod Biol. 2014 Feb;173:43-7. doi: 10.1016/j.ejogrb.2013.11.016. Epub 2013 Nov 28. PMID 24321466
- [Background] Gupta M, Emary K, Impey L. Emergency cervical cerclage: predictors of success. J Matern Fetal Neonatal Med. 2010 Jul;23(7):670-4. doi: 10.3109/14767050903387011. PMID 19883267
- [Background] Zanardini C, Pagani G, Fichera A, Prefumo F, Frusca T. Cervical cerclage in twin pregnancies. Arch Gynecol Obstet. 2013 Aug;288(2):267-71. doi: 10.1007/s00404-013-2758-3. Epub 2013 Feb 21. PMID 23430029
- [Background] Miller ES, Rajan PV, Grobman WA. Outcomes after physical examination-indicated cerclage in twin gestations. Am J Obstet Gynecol. 2014 Jul;211(1):46.e1-5. doi: 10.1016/j.ajog.2014.03.034. Epub 2014 Mar 18. PMID 24657791
- [Background] Berghella V, Roman A. Cerclage in twins: we can do better! Am J Obstet Gynecol. 2014 Jul;211(1):5-6. doi: 10.1016/j.ajog.2014.03.037. No abstract available. PMID 24972530
- [Background] Liem S, Schuit E, Hegeman M, Bais J, de Boer K, Bloemenkamp K, Brons J, Duvekot H, Bijvank BN, Franssen M, Gaugler I, de Graaf I, Oudijk M, Papatsonis D, Pernet P, Porath M, Scheepers L, Sikkema M, Sporken J, Visser H, van Wijngaarden W, Woiski M, van Pampus M, Mol BW, Bekedam D. Cervical pessaries for prevention of preterm birth in women with a multiple pregnancy (ProTWIN): a multicentre, open-label randomised controlled trial. Lancet. 2013 Oct 19;382(9901):1341-9. doi: 10.1016/S0140-6736(13)61408-7. Epub 2013 Aug 5. PMID 23924878
- [Background] Althuisius SM, Dekker GA, Hummel P, van Geijn HP; Cervical incompetence prevention randomized cerclage trial. Cervical incompetence prevention randomized cerclage trial: emergency cerclage with bed rest versus bed rest alone. Am J Obstet Gynecol. 2003 Oct;189(4):907-10. doi: 10.1067/s0002-9378(03)00718-x. PMID 14586323
- [Background] Roman A, Rochelson B, Martinelli P, Saccone G, Harris K, Zork N, Spiel M, O'Brien K, Calluzzo I, Palomares K, Rosen T, Berghella V, Fleischer A. Cerclage in twin pregnancy with dilated cervix between 16 to 24 weeks of gestation: retrospective cohort study. Am J Obstet Gynecol. 2016 Jul;215(1):98.e1-98.e11. doi: 10.1016/j.ajog.2016.01.172. Epub 2016 Jan 28. PMID 26827881
- [Derived] Roman A, Zork N, Haeri S, Schoen CN, Saccone G, Colihan S, Zelig C, Gimovsky AC, Seligman NS, Zullo F, Berghella V. Physical examination-indicated cerclage in twin pregnancy: a randomized controlled trial. Am J Obstet Gynecol. 2020 Dec;223(6):902.e1-902.e11. doi: 10.1016/j.ajog.2020.06.047. Epub 2020 Jun 25. PMID 32592693

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-02-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT02490384/Prot_SAP_000.pdf
  • Informed Consent Form (2015-05-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT02490384/ICF_001.pdf